CLINICAL TRIAL: NCT03379246
Title: Are we Supporting the Apex During Hysterectomy for Pelvic Organ Prolapse?
Brief Title: Apical Support During Hysterectomy for Pelvic Organ Prolapse
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 17-091
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-10

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective chart review using TriHealth Electronic Privacy Identification Center (EPIC) to determine whether gynecologic surgeons at a large community hospital are already meeting the recently recommended best practice of supporting the vaginal apex.

DETAILED DESCRIPTION:
The prevalence of pelvic organ prolapse (POP) in the United States is estimated to be between 40-50% with an anticipated increase over the next several decades. Approximately 300,000 women undergo surgeries to repair POP in the United States every year. Following pelvic reconstructive surgery, recurrence rates of symptomatic prolapse range between 6-30%. Our understanding of pelvic anatomy and its support has been significantly improved over recent decades, with many researchers reporting on details and mechanics previously not understood.

In November 2017, the American College of Obstetricians and Gynecologists released a new practice bulletin outlining the current standard of care for the treatment of women with pelvic organ prolapse. In this bulletin, they state that a hysterectomy alone is not adequate treatment for pelvic organ prolapse, and further that any woman having a hysterectomy for pelvic organ prolapse should undergo a concurrent apical suspension procedure as a standard of care.

The purpose of this study is to determine the proportion of patients already meeting the recently recommended best practice of supporting the vaginal apex at the time of hysterectomy for pelvic organ prolapse among the population who underwent the surgery performed at a TriHealth facility between October 2012 and October 2017.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Underwent hysterectomy for pelvic organ prolapse, performed at a TriHealth facility between October 2012 and October 2017

Exclusion Criteria:

* Age < 18 years old
* Pelvic Organ Prolapse was not an indication for their surgery
* Surgery performed by a physician of Cincinnati Urogynecology Associates.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who had hysterectomy for pelvic organ prolapse, performed by gynecologic surgeons at any of the affiliated TriHealth hospitals between October 2012 and October 2017
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catrina Crisp, MD, MSc, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hill AM, Pauls RN, Crisp CC. Practice Patterns Regarding Apical Support Procedures at Time of Hysterectomy for Pelvic Organ Prolapse. Female Pelvic Med Reconstr Surg. 2020 Dec 1;26(12):774-778. doi: 10.1097/SPV.0000000000000716. PMID 30921081

RESULTS

PARTICIPANT FLOW:
Groups:
- Pelvic Organ Prolapse: patients who underwent hysterectomy for pelvic organ prolapse at any of the affiliated TriHealth hospitals between October 2012 and October of 2017
Period: Overall Study
Arm/Group | Pelvic Organ Prolapse
Started | 236
Completed | 236
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pelvic Organ Prolapse
Number analyzed (Participants) | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.86 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 225
  African American | 7
  Asian | 1
  Multiracial | 1
  Other | 1
  Unavailable | 1
Region of Enrollment [Number; unit: participants]
  United States | 236

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Having Concurrent Apical Suspension Performed
Description: proportion of patients who had concurrent apical support procedures performed
Time Frame: at time of hysterectomy for pelvic organ prolapse
Measure: Count of Participants; unit: Participants
Arm/Group | Pelvic Organ Prolapse
Number analyzed (Participants) | 236
Participants | 66

ADVERSE EVENTS:
Time Frame: Day of surgery
Arm/Group | Pelvic Organ Prolapse
All-Cause Mortality (participants affected / at risk) | 0/236
Serious Adverse Events (participants affected / at risk) | 0/236
Other Adverse Events (participants affected / at risk) | 0/236

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT03379246/Prot_SAP_000.pdf